CLINICAL TRIAL: NCT06372132
Title: 'Treatment Outcome of Gastric Peroral Endoscopic Pyloromyotomy in Comparison With Percutaneous Endoscopic Gastrostomy With Jejunal Extension in Medically Refractory Gastroparesis: a Prospective Randomized Controlled Trial'
Brief Title: G-POEM vs PEG-J in Gastroparesis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL85305.068.23
Record Dates: First submitted 2024-02-29; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Pyloromyotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-POEM (Other)
  Interventions: Procedure: G-POEM
- PEG-J (Active Comparator)
  Interventions: Procedure: G-POEM

INTERVENTIONS:
Procedure: G-POEM — Gastric Per-Oral Endoscopic Pyloromyotomy
  Other Names: PEG J

SUMMARY:
Study design: A randomized non-blinded controlled clinical trial with two study arms (G-POEM and PEG-J). Treatment success is measured using the GCSI at baseline before intervention and six months after intervention with a possible cross-over after six months of follow-up.

Study population: 50 patients with therapy refractory GP on dietary advices, prokinetics and possibly tube feeding (gastric rest) who have already been referred for additional treatment options in the form of PEG-J/ G-POEM.

Intervention: Group 1 will receive G-POEM treatment and group 2 will receive PEG-J treatment.

Main study parameters/endpoints: A clinically meaningful treatment success six months after G-POEM treatment, measured using the GCSI-score defined as a decrease of 1 or more point.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GP
* 13C octanoic acid test or gastric scintigraphy (minimal 4-hour measurement) within the past twelve months
* 18 years old

Exclusion Criteria:

* < 18 years old
* Medical history of stomach surgery in which resection of antrum and/ or pylorus took place
* Medical history of surgical or laparoscopic pyloromyotomy
* Gastric bypass
* Current opioid use
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment success using the GCSI-score in patients with refractory GP undergoing G-POEM compared to patients receiving a PEG-J at t = 6 months. | 6 months
  A treatment success will be defined as a decrease of at least one point on the GCSI (range 0-5), representing a clinically relevant difference, six months after intervention in comparison with baseline before intervention.

SECONDARY OUTCOMES:
Number of patients with treatment success using the GCSI-score in patients with refractory GP undergoing G-POEM compared to patients receiving a PEG-J at t = 12 months. | 12 months
  We hypothesize that the treatment success rate is higher in the G-POEM group in comparison with the PEG-J intervention group twelve months after intervention compared to baseline.
Degree of quality of life using the PAGI-QOL in the G-POEM group in comparison with the PEG-J intervention six months after intervention. | 6 months
  We hypothesize that quality of life is higher in the G-POEM intervention group compared to the PEG-J intervention group six months after treatment.
Number and severity of (s)AEs in the treatment groups. | 12 months
  We hypothesize that no severe adverse events take place and the only mild to moderate adverse events that will take place are expected to be abdominal pain, pneumoperitoneum, mucosal injury, or wound infection.
Predictive value of the etiology of gastroparesis on treatment outcomes following G-POEM by measuring the rate of treatment success quantified by improvements in the GCSI-score. | 6-12 months
  We hypothesize that differences in etiology can predict treatment success after G-POEM.
Predictive value of the etiology of gastroparesis on treatment outcomes following PEG-J by measuring the rate of treatment success quantified by improvements in the GCSI-score. | 6-12 months
  We hypothesize that differences in etiology can predict treatment success after PEG-J.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Zuid-Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided